CLINICAL TRIAL: NCT02938273
Title: Bioimmunoradiotherapy (BIR) With Concurrent Avelumab, Cetuximab and Radiotherapy as First Line Treatment in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck. A Feasibility Study in Patients Unfit for Cisplatin
Brief Title: Bioimmunoradiotherapy (Cetuximab/RT/Avelumab)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N16BIR
Record Dates: First submitted 2016-09-26; First posted 2016-10-19 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — avelumab; Radiotherapy; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bioimmunoradiotherapy (Experimental): Concurrent Radiation therapy (i.e. 5 times a week, 7 weeks, total dose 70 Gy) with cetuximab (loading dose 400 mg/m2 i.v. day -7, 250 mg/m2 i.v weekly wk 1-7) and Avelumab10 mg/kg i.v. at day -7, 7, 21,35 + maintenance therapy i.e avelumab10 mg/kg i.v. every 2 weeks for 6 months (wk 8,10, 12, 14, 16, 18, 20, 22, 24, 26.
  Interventions: Drug: avelumab; Radiation: radiotherapy; Drug: cetuximab

INTERVENTIONS:
Drug: avelumab — Avelumab10 mg/kg i.v. at day -7, 7, 21,35 + maintenance therapy i.e avelumab10 mg/kg i.v. every 2 weeks for 6 months
  Other Names: MSB0010718C
Radiation: radiotherapy — 5 times a week, 7 weeks, total dose 70 Gy
Drug: cetuximab — loading dose 400 mg/m2 i.v. day -7, 250 mg/m2 i.v weekly wk 1-7
  Other Names: erbitux

SUMMARY:
This is an open-label phase IB trial with Bioimmunoradiotherapy, i.e. concurrent radiotherapy with intravenous administration of cetuximab and avelumab followed by avelumab maintenance therapy in patients with locally advanced head and neck cancer, unfit for cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be ≥18 years of age on day of signing informed consent.
* WHO Performance Status 0,1 or 2
* Have histologically confirmed Locally Advanced (i.e. stage III or IV) head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx and larynx.
* Unfit for concurrent chemoradiation with cisplatin, e.g. GFR < 60 ml/min, cardiovascular co-morbidity, hearing loss or polyneuropathy or written refusal for treatment with chemotherapy
* Be willing to provide tissue for tumor microenvironment analysis from archival tumor material (i.e. formalin fixed, paraffin embedded (FFPE) tumor tissue block not older than 42 days before start of treatment) or newly obtained core or excisional biopsy, and willingness to provide a core or excisional biopsy at day 14 (±2 days) after start of treatment.
* Have at least one measurable lesion as defined by RECIST 1.1.
* Be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Demonstrate adequate organ function, i.e. adequate bone marrow function, including:

  1. Absolute Neutrophil Count (ANC) ≥1.5 x 109/L;
  2. Platelets ≥100 x 109/L;
  3. Hemoglobin ≥6 mmol/L. Adequate renal function, i.e. estimated creatinine clearance ≥30 mL/min as calculated using the Cockcroft-Gault (CG) equation (or local institutional standard method).

Adequate liver function, including:

1. Total serum bilirubin ≤1.5 x ULN;
2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).

   * Have a negative serum pregnancy test at screening (for females of childbearing potential).
   * Both male and female subjects should agree to use highly effective contraception if the risk of conception exists. (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential and men able to father a child must agree to use 2 highly effective contraception, defined as methods with a failure rate of less than 1 % per year.) Highly effective contraception is required throughout the study and for at least 120 days after Avelumab treatment.

Exclusion Criteria:

- Prior treatment with: Systemic therapy, radiotherapy or surgery directed at locally advanced SCCHN. Immunotherapy with IL-2, IFN-α, or anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.

* A diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Current or prior use of immunosuppressive medication within 7 days prior to registration, except the following:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra-articular injection);
  * Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥3), any history of anaphylaxis, or uncontrolled asthma (i.e., 3 or more features of partially controlled asthma Global Initiative for Asthma 2011.
* Known prior or suspected hypersensitivity to study drugs or any component in their formulations.
* Diagnosis of any other malignancy within 5 years prior to start of treatment except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix, or low-grade (Gleason 6 or below) prostate cancer on surveillance with no plans for treatment intervention (e.g. surgery, radiation, or castration).
* Significant acute or chronic infections including, among others:

  * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
  * Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive)
* Prior organ transplantation, including allogeneic stem cell transplantation
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent, except the following:

  1. Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment
  2. Subjects requiring hormone replacement with corticosteroids if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
  3. Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation)
* Persisting toxicity related to prior therapy of Grade >1; however, alopecia and sensory neuropathy Grade ≤ 2 is acceptable
* Pregnancy or lactation
* Known alcohol or drug abuse
* All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated influenza vaccines).
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, deep vein thrombosis or symptomatic pulmonary embolism.
* Subjects with brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
occurence of grade 3-5 toxicity in new combination | 6 months after start of treatment
  according to CTC 4.03

SECONDARY OUTCOMES:
Overall Response Rate | at week 10 and week 26 of treatment

OTHER OUTCOMES:
differences in tumor microenvironment | prior to treatment and at day 14
  investigate therapy induced changes in tumor microenvironment in tissue biopsies through immunochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul de Boer, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elbers JBW, Al-Mamgani A, Tesseslaar MET, van den Brekel MWM, Lange CAH, van der Wal JE, Verheij M, Zuur CL, de Boer JP. Immuno-radiotherapy with cetuximab and avelumab for advanced stage head and neck squamous cell carcinoma: Results from a phase-I trial. Radiother Oncol. 2020 Jan;142:79-84. doi: 10.1016/j.radonc.2019.08.007. Epub 2019 Sep 26. PMID 31563412